CLINICAL TRIAL: NCT00752219
Title: A Prospective, Multicenter, Double-blind, Randomized, Comparative Study to Estimate the Safety, Tolerability and Efficacy of NXL104/Ceftazidime Plus Metronidazole vs. Meropenem in the Treatment of Complicated Intra-abdominal Infections in Hospitalized Adults
Brief Title: Prospective Multicenter Doubleblind Randomized Study of NXL104/Ceftazidime + Metronidazole vs. Meropenem in Treatment of Complicated Intra-abdominal Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NXL-104/2002; C3591014 (Other: Alias Study Number)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Complicated Intra-abdominal Infections
MeSH Terms: interventions — Ceftazidime; avibactam; Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NXL104/CAZ/MTZ (Experimental): NXL104/ceftazidime + metronidazole
  Interventions: Drug: ceftazidime/NXL104 + metronidazole
- Meropenem (Active Comparator)
  Interventions: Drug: meropenem

INTERVENTIONS:
Drug: ceftazidime/NXL104 + metronidazole — IV TID
  Arms: NXL104/CAZ/MTZ
Drug: meropenem — IV TID
  Other Names: merrem
  Arms: Meropenem

SUMMARY:
The purpose of this study is to determine whether NXL104 plus ceftazidime is effective in the treatment of complicated intra-abdominal infections as compared to a comparator group.

ELIGIBILITY:
Inclusion Criteria:

* complicated intra-abdominal infections

Exclusion Criteria:

* infections limited to hollow viscus
* ischemic bowel disease without perforation
* acute suppurative cholangitis
* acute necrotizing pancreatitis
* pts to undergo stated abdominal repair, open abdomen technique or marsupialization
* Apache II >25

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-03-31 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center Dept of Surgery, Los Angeles, California
  - Michael S. Somero Research Division, Palm Springs, California
  - Henry Ford Health System, Detroit, Michigan
  - Mercury Street Medical Group, Butte, Montana
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Summa Health Systems, Akron, Ohio
  - Remington-Daviss Inc, Columbus, Ohio
  - ID Clinical Research Ltd, Toledo, Ohio
- Bulgaria (5):
  - UMHAT Sveti Georgi 3rd Clinical of Surgery, Plovdiv
  - MHAT Rousse, 2nd Clinical of Surgery, Rousse
  - CCB Ministry of Interior Clinical of Surgery, Sofia
  - Multiprofile Hospital for Active Trt Emergency Med, Sofia
  - UMHAT Queen Joanna-ISUL, Clinical of Surgery, Sofia
- France (3):
  - Hospital Saint Joseph Marseille, Marseille
  - Hospital L'Archet II, Nice
  - CHU Nimes, Nîmes
- India (8):
  - Medisurge Hospital Ahmedabad, Ahmedabad
  - Medisys Clinisearch India Pvt Ltd, Bangalore
  - MS Ramaiah Memorial Hospital Bangalore, Bangalore
  - Victoria Hospital Bangalore, Bangalore
  - Suyash Hospital Indore, Indore
  - SR Kalla General and Gastro Hospital, Jaipur
  - Amrita Institute of Medical Sciences, Cochin, Kochi
  - Lucknow Cancer Institute Lucknow, Lucknow
- Lebanon (5):
  - Al-Zahraa university Hospital, Beirut
  - Makassed General Hospital, Beirut
  - Rafik Heriri University Hospital, Beirut
  - Hammound Hospital University Medical Center, Saida
  - Labib Medical Center, Saida
- Poland (5):
  - Slaski Uniwersytet Medyczny, Katowice
  - Pomorskie Centrum Traumatologii, Nowe Ogrody
  - Katedra i Klinika Chirurgii Ogolnej, Warsaw
  - Samodzielny Publiczny, Warsaw
  - Akademicki Szpital Kliniczn, Wroclaw
- Romania (4):
  - Coltea Clinical Hospital, Bucharest
  - Floreasca Clinical Emergency Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - University Emergency Hospital Bucharest, Bucharest
- Russia (6):
  - City Clinical Hospital # 13, Moscow
  - City Clinical Hospital # 1, Moscow
  - FGU National Medical Surgery, Moscow
  - Moscow City Clinical Hospital # 31, Moscow
  - SMO of Clinical Trials, Smolensk
  - North-Ossetian Medical Academy, Vladikavkas

REFERENCES:
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279

RESULTS

PARTICIPANT FLOW:
Groups:
- NXL104/Ceftazidime + Metronidazole: Participants received intravenous dose of 500 milligram (mg) of NXL104, 2000 mg of ceftazidime and 500 mg of metronidazole every 8 hour, for up to a maximum duration of 14 days. Participants were followed up to a maximum of 6 weeks post therapy.
- Meropenem: Participants received intravenous dose of 1000 mg of meropenem every 8 hour, for up to a maximum duration of 14 days. Participants were followed up to a maximum of 6 weeks post therapy.
Period: Overall Study
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Started | 102 | 102
Treated | 101 | 102
Completed | 91 | 96
Not Completed | 11 | 6
Not completed — Clinical failure | 0 | 1
Not completed — Adverse Event | 5 | 3
Not completed — Protocol deviation | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Randomized but not treated | 1 | 0
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 43.0 (15.93) | 42.6 (18.09) | 42.8 (17.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at informed consent
  Participants
    Female | 31 | 21 | 52
    Male | 70 | 81 | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at the Test of Cure (TOC) Visit
Description: Clinical response was defined as complete resolution or significant improvement of signs and symptoms of the index infection. No further antimicrobial therapy or surgical or radiological intervention was required. This clinical response was measured in participants who were microbiologically evaluable (ME) at baseline.
Time Frame: Test of cure visit: 2 weeks post-therapy (Day 28)
Population: ME set:clinically evaluable(CE)subset with atleast 1 etiologic pathogen isolated from a clinically relevant specimen in initial culture susceptible in both study agents. CE set:participants diagnosed with intraperitoneal infection confirmed by operative findings with adequate therapy and information to determine clinical outcome at specified visit.
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 62 | 71

2. Secondary Outcome: Number of Participants With Clinical Response at the End of Intravenous (IV) Therapy
Description: Clinical response was defined as complete resolution or significant improvement of signs and symptoms of the index infection. No further antimicrobial therapy or surgical or radiological intervention was required. This clinical response was measured in participants who were ME at baseline.
Time Frame: End of IV therapy: From Day 5 to Day 14
Population: ME population: A subset of CE population with at least 1 etiologic pathogen isolated from a clinically relevant specimen in initial culture susceptible in both study agents.
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 66 | 74

3. Secondary Outcome: Number of Participants With Clinical Response at the Late Follow-up Visit
Description: as for outcome 2
Time Frame: Late follow-up visit: 4 to 6 weeks post-therapy (up to 8 weeks)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 62 | 71

4. Secondary Outcome: Number of Participants With Microbiological Response at the Test of Cure Visit
Description: Microbiological response was defined as eradication of pathogen identified (absence of causative pathogens from appropriately obtained specimens at site of infection) or presumptive eradication of pathogens (absence of material to culture in a participant who had responded clinically to treatment). This clinical response was measured in participants who were ME at baseline.
Time Frame: Test of cure visit: 2 weeks post-therapy (Day 28)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 62 | 71

5. Secondary Outcome: Number of Participants With Microbiological Response at the End of IV Therapy
Description: as for outcome 4
Time Frame: End of IV therapy: From Day 5 to Day 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 66 | 74

6. Secondary Outcome: Number of Participants With Microbiological Response at the Late Follow-up Visit
Description: Favorable: eradication (absence of causative pathogens from appropriately obtained specimens at site of infection) or presumptive eradication (absence of material to culture in a patient who had responded clinically to treatment)
Time Frame: Late follow-up visit: 4 to 6 weeks post-therapy (up to 8 weeks)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 68 | 76
participants | 62 | 71

7. Secondary Outcome: Number of Participants With Clinical Response in Clinically Evaluable (CE) Participants at the Test of Cure Visit
Description: Clinical response was defined as complete resolution or significant improvement of signs and symptoms of the index infection. No further antimicrobial therapy or surgical or radiological intervention was required.
Time Frame: Test of cure visit: 2 weeks post-therapy (Day 28)
Population: CE population included all randomized participants diagnosed with intraperitoneal infection confirmed by operative findings, received adequate therapy and had information to determine clinical outcome at specified visit.
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 87 | 90
participants | 80 | 85

8. Secondary Outcome: Number of Participants With Clinical Response in CE Participants at the End of IV Therapy
Description: as for outcome 7
Time Frame: End of IV therapy: From Day 5 to Day 14
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 87 | 89
participants | 84 | 87

9. Secondary Outcome: Number of Participants With Clinical Response in CE Participants at the Late Follow-up Visit
Description: as for outcome 7
Time Frame: Late follow-up visit: 4 to 6 weeks post-therapy (up to 8 weeks)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 86 | 89
participants | 79 | 84

10. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 6 weeks after last dose of study treatment that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 6 weeks after last dose of study treatment (up to a maximum of 8 weeks)
Population: Safety population included all participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Number analyzed (Participants) | 101 | 102
participants
  AEs | 65 | 59
  SAEs | 9 | 11

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | NXL104/Ceftazidime + Metronidazole | Meropenem
Serious Adverse Events (participants affected / at risk) | 9/101 | 11/102
Other Adverse Events (participants affected / at risk) | 41/101 | 36/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NXL104/Ceftazidime + Metronidazole (N=101) | Meropenem (N=102)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Gastric Perforation (Gastrointestinal disorders) | 1 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Multi-Organ Failure (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Postoperative Abscess (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 0 | 1
Hepatic Enzyme Increased (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Injury, poisoning and procedural complications) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheo-Oesophageal Fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NXL104/Ceftazidime + Metronidazole (N=101) | Meropenem (N=102)
Vomiting (Gastrointestinal disorders) | 14 | 5
Nausea (Gastrointestinal disorders) | 10 | 6
Abdominal Pain (Gastrointestinal disorders) | 8 | 3
Pyrexia (General disorders) | 9 | 11
Aspartate Aminotransferase Increased (General disorders) | 9 | 15
Alanine Aminotransferase Increased (General disorders) | 8 | 13
Blood Alkaline Phosphatase Increased (General disorders) | 9 | 7
Platelet Count Increased (General disorders) | 4 | 7
White Blood Cell Count Increased (General disorders) | 5 | 6
Haematuria (Renal and urinary disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.